CLINICAL TRIAL: NCT05226429
Title: Safety and Immunogenicity of UNAIR Inactivated COVID-19 Vaccine in Healthy Populations Aged 18 Years and Above (Phase I/II)
Brief Title: UNAIR Inactivated COVID-19 Vaccine
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr. Soetomo General Hospital (Other Government)
Collaborators: Indonesia-MoH (Other Government); Universitas Airlangga (Other); Bioxis Pharmaceuticalls (Industry)
Responsible Party: Principal Investigator, Dr. Dominicus Husada, dr., DTM&H, MCTM(TP), Sp.A(K), Vice Chair of Institutional Review Board, Dr. Soetomo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UNAIR-MP-INAKTIF-001
Record Dates: First submitted 2022-01-20; First posted 2022-02-07 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: COVID-19 Pandemic; Vaccine Reaction
Keywords: Inactivated COVID-19 Vaccine; Immunogenicity; Indonesia; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: There will be 3 groups in phase I. Two adult groups (18 year old and above) with two different doses (3 and 5 μg) and 1 control group using Coronavac-BioFarma vaccine. There will be the same 3 groups in phase II. Two treatment groups of adult will use 2 kind of doses as in phase I. The other group is for control (Coronavac-BioFarma vaccine). The vaccines will be administered with 2-dose schedule, intramuscularly. All cohorts will be followed for 12 months.
Who Masked: Participant, Investigator
Masking Description: In this clinical trial, the experimental vaccine and the control vaccine will have different packages. In order to maintain the blinding process, the unblinded team will be appointed to place the vaccine in the syringe. The injection team (other team members) will later inject the vaccines according to the random group that has been selected. The unblinded team consists mostly of pharmacists and they will also have responsibilities to taking care of the vaccines and all of related documents. The injection team does not know what kind of vaccine is in the syringe. The injection team is also different from the observer team (those who will observe the subjects after the injection). This observer team does not know what kind of vaccine that already be given to the subjects.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- UNAIR Inactivated COVID-19 Vaccine 3 microgram (Experimental)
  Interventions: Biological: UNAIR Inactivated COVID-19 Vaccine
- UNAIR Inactivated COVID-19 Vaccine 5 microgram (Experimental)
  Interventions: Biological: UNAIR Inactivated COVID-19 Vaccine
- CoronaVac Biofarma COVID-19 Vaccine (Active Comparator)
  Interventions: Biological: CoronaVac Biofarma COVID-19 Vaccine

INTERVENTIONS:
Biological: UNAIR Inactivated COVID-19 Vaccine — UNAIR Inactivated Covid-19 Vaccine contains S protein of SARS-CoV-2 virus, Aluminium hydroxide gel, 10 mM L-Histidine buffer, 0.005% Tween Polysorbate 80, and 0.9% Sodium chloride. Vaccine will be prepared in vial (1 ml per vial). One vial will be used for one injection only. The vial should be shaken well before injection.
  Arms: UNAIR Inactivated COVID-19 Vaccine 3 microgram; UNAIR Inactivated COVID-19 Vaccine 5 microgram
Biological: CoronaVac Biofarma COVID-19 Vaccine — Control vaccine in this study is existing CoronaVac-BioFarma inactivated COVID-19 vaccine which has been used widely in Indonesia.
  Arms: CoronaVac Biofarma COVID-19 Vaccine

SUMMARY:
This is a randomized, observer blind, controlled phase I/II study to evaluate the Safety, Reactogenicity, and Immunogenicity of UNAIR Inactivated Covid-19 Vaccine in Healthy Populations Aged 18 Years and Above. UNAIR Inactivated Covid-19 Vaccine is an inactivated vaccine developed by Airlangga University (Universitas Airlangga / UNAIR) made of SARS-CoV-2 virus isolated from a patient in Surabaya, Indonesia, composed with aluminium hydroxy gel, tween 80, and L-histidine. This study will be the first in human.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults and elderly, males and females, 18 years of age and above. Healthy status will be determined by the investigator based on medical history, clinical laboratory results, vital sign measurements, and physical examination at screening.
2. Subjects have been informed properly regarding the study and signed the informed consent form
3. Subject will commit to comply with the instructions of the investigator and the schedule of the trial
4. Female subjects of childbearing potential must agree to consistently use any methods of contraception (except the periodic abstinence) from at least 21 days prior to enrollment and through 6 months after the last vaccination.
5. Participants agree not to donate bone marrow, blood, and blood products from the first study vaccine administration until 3 months after receiving the last dose of study vaccine.
6. Participants must be willing to provide verifiable identification, has means to be contacted and to contact the investigator during the study.

Exclusion Criteria:

1. Subjects concomitantly enrolled or scheduled to be enrolled in another trial.
2. Evolving mild, moderate, and severe illness, especially infectious diseases or fever (axillary temperature 37.5 degree Celcius or more) concurrent or within 7 days prior to first study vaccination. This includes respiratory or constitutional symptoms consistent with SARS-CoV-2 (cough, sore throat, difficulty in breathing, etc)
3. Known history of allergy to any component of the vaccines
4. History of uncontrolled coagulopathy or blood disorders contraindicating intramuscular injection
5. Any autoimmune or immunodeficiency disease/condition
6. Subjects who has received in the previous 4 weeks a treatment likely to alter the immune response (intravenous immunoglobulin, blood derived products, long term corticosteroid - more than 2 weeks, and so on), OR anticipation of the need for immunosuppressive treatment within 6 months after last vaccination. The use of topical or nasal steroid will be permitted. Inhaled glucocorticoids is prohibited.
7. Chronic disease, inclusive of uncontrolled hypertension, congestive heart failure, chronic obstructive pulmonary disease, asthma, chronic urticaria, diabetes requiring use of medicine
8. Any abnormality or chronic disease which according to the investigator might interfere with the assessment of the trial objectives
9. Individuals who previously receive any vaccines against Covid-19
10. Subjects already immunized with any vaccine within 4 weeks prior and expect to receive other vaccines within 60 days following the first dose
11. Individuals who have a previously ascertained Covid-19 in the period of 3 months before the first recruit of this study, or in a close contact in the last 14 days with confirmed case of Covid-19
12. Positive test for SARS-CoV-2 (Antigen or PCR) at screening prior to first vaccination. Testing may be repeated during the screening period if exposure to positive confirmed case of SARS-CoV-2 is suspected, at the discretion of investigator.
13. History of alcohol or substance abuse
14. HIV patients.
15. Malignancy patients within 5 years prior to first study vaccination.
16. Any neurological disease or history of significant neurological disorder such as meningitis, encephalitis, Guillain-Barre Syndrome, multiple sclerosis, etc
17. Vital sign abnormalities and clinical laboratory abnormalities as decided by the investigators. Vital sign measurements and clinical laboratory testing may be repeated before the final decision.
18. Women who are pregnant, breastfeeding, or who plan to become pregnant during the study.
19. Participant has major psychiatric problem or illness
20. Participant cannot communicate reliably with the investigator
21. Participant has contraindication to intramuscular injection and blood draws, such as bleeding disorders or phobia.
22. Participant had major surgery within 12 weeks before vaccination which will not be fully recovered, or has major surgery planned during the time participant is expected to participate in the study or within 6 months after the last dose of study vaccine administration.
23. Any condition that in the opinion of the investigators would pose a health risk to the subject if enrolled or could interfere with the evaluation of the vaccine or interpretation of the study results
24. Study team members.
25. Subject planning to move from the study area before the end of study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 495 (Estimated)
Dates: Start 2022-02-08 (Actual); Primary Completion 2023-04-06 (Actual); Study Completion 2023-07-06 (Estimated)

PRIMARY OUTCOMES:
Solicited clinical (local and systemic), laboratory, and unsolicited adverse events | 7 days each vaccination
  The number of adverse events occur among participants.
Solicited clinical (local and systemic), laboratory, and unsolicited adverse events | 28 days after each vaccination
  The number of adverse events occur among participants.
SARS-CoV-2 neutralization antibodies | 28 days after the second vaccination
  The level of SARS-CoV-2 neutralization antibodies in participants.
SARS-CoV-2 binding antibodies | 28 days after the second vaccination
  The level of SARS-CoV-2 binding antibodies in participants.
Th1 and Th2 | 28 days after the second vaccination
  Th1 and Th2 levels in participants.

SECONDARY OUTCOMES:
Solicited clinical (local and systemic), laboratory, and unsolicited adverse events | 3, 6, and 12 months after the first vaccination
  The number of adverse events occur among participants.
SARS-CoV-2 neutralization antibodies | 3, 6, and 12 months after the first vaccination
  The level of SARS-CoV-2 neutralization antibodies in participants.
SARS-CoV-2 binding antibodies | 3, 6, and 12 months after the first vaccination
  The level of SARS-CoV-2 binding antibodies in participants.
Th1 and Th2 | 3, 6, and 12 months after the first vaccination
  Th1 and Th2 levels in participants.

CONTACTS AND LOCATIONS:
Overall Officials: Dominicus Husada, MD, Principal Investigator — Dr. Soetomo General Hospital
Locations (1):
- Dr. Soetomo General Hospital, Surabaya, East Java, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided
There is not yet plan to share IPD with other researchers.